CLINICAL TRIAL: NCT06354504
Title: Gingival Crevicular Fluid (GCF) Bactericidal/Permeability-increasing Protein (BPI) and Interleukin (IL)-1beta in Periodontitis Patients: Non-surgical Periodontal Treatment Effects
Brief Title: Bactericidal Permeability Protein Inhibitor and Interleukin-1beta Levels After Non-surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nezahat Arzu Kayar, Clinical Professor, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.02.2019/177
Record Dates: First submitted 2024-03-07; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healty (Experimental): Non-surgical periodontal treatment
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Scaling and root planing in two sessions over the course of a 48-hour period comprised the standard treatment procedure

SUMMARY:
The aim of this study was to examine the relationship between healing response after non-surgical periodontal treatment and baseline gingival crevicular fluid (GCF) levels of bactericidal/permeability-increasing protein (BPI) and interleukin-1beta (IL-1ß).

DETAILED DESCRIPTION:
Bactericidal/permeability-increasing proteins (BPI) specific and powerful effect against Gram negative bacteria and their LPSs is completely observable in biological fluids such as plasma, serum, and whole blood.

Objective: It is the evaluation of periodontal disease effect of BPI and interleukin-1 beta (IL-1 β) levels in gingival fluid before and after non-surgical periodontal treatment (NSPT)in patients with periodontal disease.

Method: Thirty systemically healthy and non-smoking individuals with periodontitis were included in the study. Before NSPT, the clinical parameters of plaque index (PI), gingival index (GI), probing depth (PD), clinical attachment level (CAS), bleeding on probing (BOP) were measured. The gingival fluid samples were taken using the paper strip method. The same procedures were repeated at 6 weeks and 6 months after non-surgical periodontal treatment. ELISA method was used for the analysis of the samples

ELIGIBILITY:
Inclusion Criteria

Systemically healthy,

* Stage II or III, Grade A periodontitis
* Having at least 20 permanent teeth (excluding third molars and any tooth loss induced by -non-periodontal causes).

Exclusion Criteria:

Smoking,

* use of alcohol; pregnancy or lactation; intake ofantibiotics, steroidal or non-steroidal anti-inflammatory drugs within the last 6 months
* having received periodontal treatment within the last 6 months

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid Bactericidal/permeability-increasing proteins levels | through study completion, an average of 1 year
  Gingival Crevicular Fluid Bactericidal Permeability Increasing Protein levels in periodonitis patients after Non-surgical periodontal treatment

SECONDARY OUTCOMES:
Gingival crevicular fluid interleukin-1Beta levels | through study completion, an average of 1 year
  Gingival Crevicular Fluid IL-1β in periodonitis patients after Non-surgical periodontal treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz Üniversity, Antalya
  - Akdeniz Üniversitesi Diş Hekimliği Fakültesi, Antalya

IPD SHARING:
Plan to Share IPD: No